CLINICAL TRIAL: NCT07159581
Title: Evaluation of the Effect of Gene Therapy for Wilson Disease With 64CuCl₂ PET Imaging
Brief Title: Gene Therapy for Wilson Disease Evaluated by 64Cu PET/CT
Status: Enrolling by invitation | Type: Observational
Sponsor: Thomas Damgaard Sandahl (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Thomas Damgaard Sandahl, Consultant, MD, PhD, University of Aarhus
Organization: University of Aarhus (Other)
Other Study IDs: 1-10-72-146-24
Record Dates: First submitted 2025-08-22; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Wilson Disease
Keywords: positron emission tomography; 64Cu; wilson disease; gene therapy; copper metabolism
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wilson disease patients: UX701

SUMMARY:
The primary objective of this study is to investigate the effect of gene therapy (UX704) on copper distribution and excretion in Wilson disease patients. The effect is investigated using 64Cu positron emission tomography scans combined with a CT scan.

DETAILED DESCRIPTION:
Patients entering this study are included from the ongoing clinical study "A Phase 1/ 2/ 3 Study of UX701 Gene Therapy in Adults With Wilson Disease" (NCT04884815). The patients will have received gene therapy as part of the clinical study. This study is an extension study that aims to specifically monitor the effect of gene therapy on copper distribution and excretion using 64Cu PET/CT.

Patients will receive 40-80 MBq 64CuCl2 intravenously and will undergo three PET/CT scans during the next 20 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Wilson disease who have received gene therapy (UX701) as part of NCT04884815
* Age above 18 years
* Women of childbearing potential must accept to use safe contraception at the time of the PET scans: Spiral or hormonal contraception (oral pills, implants, transdermal patches, vaginal rings, or depot injections)
* At the day of the first PET scan, a negative urine pregnancy test is required for women of childbearing potential
* Before the first PET scan, a signed informed consent must be completed

Exclusion Criteria:

* Known hypersensitivity to Cu-64, copper in general, or other components of the radiotracer formulation
* Claustrophobia
* Pregnancy, breastfeeding, or plans to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Wilson disease who have received gene therapy (UX701) as part of NCT04884815 are referred by the primary investigator of NCT04884815 to participate in this study. If they fulfil other eligibility criteria, they are invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Ratio of liver SUV at 20 hours to liver SUV at 1 hours after injection of Cu64 | From first to last scan
  The liver SUV is measured as the mean of five spherical VOIs (20 mm in diameter) placed in the right liver lobe, with distance to the organ borders and large blood vessels. The ratio is a measure of whether the tracer is retained in the liver (ratio > 1) or is excreted from the liver (ratio < 1).

SECONDARY OUTCOMES:
Gallbladder SUV at 1 hour, 6 hours and 20 hours after injection of 64Cu | From first to last scan
  SUV in a VOI covering the entire gallbladder
Percentage of injected dose in the blood at 1 hour, 6 hours and 20 hours after injection of 64Cu | From first to last scan
  Radioactivity in the blood is measured by placing a cylindrical VOI in the descending aorta. From this VOI, the kilobecquerel/ml is found. The percentage of injected dose is found by correcting for decay and multiplying by the organ volume (estimated blood volume 5% of body weight, and the density of blood is 1 g/ml).

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared in order to safeguard patient privacy. Group data will be available upon reasonable request after publication of the results.

REFERENCES:
- [Background] Kirk FT, Munk DE, Swenson ES, Quicquaro AM, Vendelbo MH, Larsen A, Schilsky ML, Ott P, Sandahl TD. Effects of tetrathiomolybdate on copper metabolism in healthy volunteers and in patients with Wilson disease. J Hepatol. 2024 Apr;80(4):586-595. doi: 10.1016/j.jhep.2023.11.023. Epub 2023 Dec 10. PMID 38081365
- [Background] Sandahl TD, Gormsen LC, Kjaergaard K, Vendelbo MH, Munk DE, Munk OL, Bender D, Keiding S, Vase KH, Frisch K, Vilstrup H, Ott P. The pathophysiology of Wilson's disease visualized: A human 64 Cu PET study. Hepatology. 2022 Jun;75(6):1461-1470. doi: 10.1002/hep.32238. Epub 2022 Jan 10. PMID 34773664